CLINICAL TRIAL: NCT04940364
Title: An Open-Label Parallel-Dose Study of the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Single Doses of Subcutaneously and Intravenously Administered Pozelimab as Monotherapy and in Combination With Single Doses of Subcutaneously Administered Cemdisiran in Japanese Healthy Volunteers
Brief Title: A Study to Examine the Safety, Tolerability and Biological Effects of Single Doses of Subcutaneously and Intravenously Administered Pozelimab as Monotherapy and in Combination With Single Doses of Subcutaneously Administered Cemdisiran in Adult Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3918-HV-20117; 2021-001794-23 (EudraCT Number)
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Pozelimab: Single-dose SC on day 1
  Interventions: Drug: Pozelimab
- Cohort 2 (Experimental): Pozelimab: Single-dose IV on day 1
  Interventions: Drug: Pozelimab
- Cohort 3 (Experimental): Pozelimab: Single-dose SC on day 29 Cemdisiran: Single-dose SC on day 1
  Interventions: Drug: Pozelimab; Drug: Cemdisiran
- Cohort 4 (Experimental): Pozelimab: Single-dose SC on day 1 Cemdisiran: Single-dose SC on day 1
  Interventions: Drug: Pozelimab; Drug: Cemdisiran
- Cohort 5 (Experimental): Optional Pozelimab: Single-dose SC on day 1 or day 29 Cemdisiran: Single-dose SC on day 1
  Interventions: Drug: Pozelimab; Drug: Cemdisiran
- Cohort 6 (Experimental): Pozelimab: Single-dose IV on day 1
  Interventions: Drug: Pozelimab

INTERVENTIONS:
Drug: Pozelimab — Administered intravenous (IV) or subcutaneous (SC) per protocol
  Other Names: REGN3918
Drug: Cemdisiran — Administered SC per protocol
  Other Names: ALN-CC5
  Arms: Cohort 3; Cohort 4; Cohort 5

SUMMARY:
The primary objective of the study is to assess the concentration-time profiles of total pozelimab, total C5, cemdisiran, and cemdisiran metabolite(s) in Japanese adult participants following single doses of intravenous (IV) and subcutaneous (SC) pozelimab and SC cemdisiran when administered on the same day or sequentially 28 days apart.

The secondary objectives of the study are:

* To evaluate the safety and tolerability of pozelimab alone and in combination with cemdisiran in healthy Japanese adult participants
* To assess the pharmacodynamic (PD) profile of pozelimab alone and in combination with cemdisiran in healthy Japanese adult participants
* To assess the immunogenicity of pozelimab and cemdisiran in healthy Japanese adult participants

ELIGIBILITY:
Key Inclusion Criteria:

1. Japanese participant must be:

   1. Be Japanese, born in Japan, and have both biologic parents and 4 biologic grandparents who are ethnically Japanese and born in Japan
   2. Have maintained a Japanese lifestyle, with no significant change since leaving Japan, including having access to Japanese food and adhering to a Japanese diet
   3. Living < 10 years outside of Japan
2. Has a Body Mass Index (BMI) between 18 and 30 kg/m2 (inclusive) at screening visit
3. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and ECGs performed at screening and/or prior to administration of initial dose of study drug
4. Is in good health based on laboratory safety testing obtained at the screening visit Note: Participant with suspected or confirmed Gilbert's disease can be enrolled in the study
5. Willing to undergo vaccination against N. meningitidis unless participant has documentation of completed series of vaccinations within the past 2 years of the screening visit
6. Must have two consecutive negative COVID-19 tests at least 48 hours apart and within 7 days prior to study drug administration Note: The test may be the point of care quantitative reverse transcriptase polymerase chain reaction (RT-qPCR) test or approved COVID-19 antigen test at the discretion of the investigator.

Key Exclusion Criteria:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease, as assessed by the investigator as defined in the protocol
2. Presents any concern to the study investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
3. Hospitalization (>24 hour) for any reason within 30 days of the screening visit
4. Has a confirmed positive drug test result at the screening visit and/or prior to enrollment; or a history of alcohol and/or drug abuse within a year prior to the screening visit
5. Is positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) at the screening visit
6. Is positive for hepatitis C antibody and positive for qualitative (i.e., detected) hepatitis C virus (HCV) RNA test at the screening visit
7. Within the previous 2 months of the screening visit has a history of bacterial, protozoal, viral or parasite infection (including COVID-19) and/or persistent chronic or active recurring infection which require treatment with antibiotics, antivirals, or antifungals
8. Known or suspected COVID-19 disease at screening and/or prior to 1st dose administration

NOTE: Other protocol-defined Inclusion and Exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Concentrations of pozelimab in serum over time | Up to 20 weeks
Concentrations of cemdisiran in plasma over time. | Up to 20 weeks

SECONDARY OUTCOMES:
The incidence and severity of treatment-emergent adverse events (TEAE) in subjects administered pozelimab with/without cemdisiran | Up to 20 weeks
Concentrations of total C5 in plasma over time | Up to 20 weeks
Change from baseline in CH50 over time | Up to 20 weeks
Incidence of treatment-emergent anti-drug antibodies (ADA) to pozelimab | Up to 20 weeks
Incidence of treatment-emergent ADA to cemdisiran | Up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/